CLINICAL TRIAL: NCT01443169
Title: A Phase 1, Randomized, Open Label, Single Dose, 5-treatment, 5- Period Crossover Study in Healthy Volunteers to Assess The Safety, Tolerability, and Pharmacokinetics of Four Controlled Release Pregabalin Tablet Formulations Administered Following an Evening Meal and the Immediate Release Formulation Administered Fasted
Brief Title: A 5-treatment, Study in Healthy Volunteers to Assess The Safety, Tolerability, and Pharmacokinetics of Four Controlled Release (CR) Pregabalin Tablet Formulations and the Immediate Release (IR) Formulation Administered Fasted
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0081286
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Pharmacokinetic; relative oral bioavailability; pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental)
  Interventions: Drug: Sequence 1 - Treatment A: Controlled Release Pregabalin; Drug: Sequence 1 - Treatment B: Controlled Release Pregabalin; Drug: Sequence 1 - Treatment C:Controlled Release Pregabalin; Drug: Sequence 1 - Treatment D: Controlled Release Pregabalin; Drug: Sequence 1 - Treatment E: Immediate Release Pregabalin
- Sequence 2 (Experimental)
  Interventions: Drug: Sequence 2 - Treatment B: Controlled Release Pregabalin; Drug: Sequence 2 - Treatment D: Controlled Release Pregabalin; Drug: Sequence 2 - Treatment A: Controlled Release Pregabalin; Drug: Sequence 2 - Treatment C: Controlled Release Pregabalin; Drug: Sequence 2 - Treatment E: Immediate Release Pregabalin
- Sequence 3 (Experimental)
  Interventions: Drug: Sequence 3 - Treatment C: Controlled Release Pregabalin; Drug: Sequence 3 - Treatment A: Controlled Release Pregabalin; Drug: Sequence 3 - Treatment D: Controlled Release Pregabalin; Drug: Sequence 3 - Treatment B: Controlled Release Pregabalin; Drug: Sequence 3 - Treatment E: Immediate Release Pregabalin
- Sequence 4 (Experimental)
  Interventions: Drug: Sequence 4 - Treatment D: Controlled Release Pregabalin; Drug: Sequence 4 - Treatment C: Controlled Release Pregabalin; Drug: Sequence 4 - Treatment B: Controlled Release Pregabalin; Drug: Sequence 4 - Treatment A: Controlled Release Pregabalin; Drug: Sequence 4 - Treatment E: Immediate Release Pregabalin

INTERVENTIONS:
Drug: Sequence 1 - Treatment A: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, heavier tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 1
Drug: Sequence 1 - Treatment B: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 1
Drug: Sequence 1 - Treatment C:Controlled Release Pregabalin — 330 mg CR tablet (slow dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 1
Drug: Sequence 1 - Treatment D: Controlled Release Pregabalin — 330 mg CR reference tablet administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 1
Drug: Sequence 1 - Treatment E: Immediate Release Pregabalin — 300 mg IR capsule administered in the evening in the fasted state.
  Arms: Sequence 1
Drug: Sequence 2 - Treatment B: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 2
Drug: Sequence 2 - Treatment D: Controlled Release Pregabalin — 330 mg CR reference tablet administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 2
Drug: Sequence 2 - Treatment A: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, heavier tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 2
Drug: Sequence 2 - Treatment C: Controlled Release Pregabalin — 330 mg CR tablet (slow dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 2
Drug: Sequence 2 - Treatment E: Immediate Release Pregabalin — 300 mg IR capsule administered in the evening in the fasted state.
  Arms: Sequence 2
Drug: Sequence 3 - Treatment C: Controlled Release Pregabalin — 330 mg CR tablet (slow dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 3
Drug: Sequence 3 - Treatment A: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, heavier tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 3
Drug: Sequence 3 - Treatment D: Controlled Release Pregabalin — 330 mg CR reference tablet administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 3
Drug: Sequence 3 - Treatment B: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 3
Drug: Sequence 3 - Treatment E: Immediate Release Pregabalin — 300 mg IR capsule administered in the evening in the fasted state.
  Arms: Sequence 3
Drug: Sequence 4 - Treatment D: Controlled Release Pregabalin — 330 mg CR reference tablet administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 4
Drug: Sequence 4 - Treatment C: Controlled Release Pregabalin — 330 mg CR tablet (slow dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 4
Drug: Sequence 4 - Treatment B: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, lighter tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 4
Drug: Sequence 4 - Treatment A: Controlled Release Pregabalin — 330 mg CR tablet (fast dissolution, heavier tablet) administered after a 600 to 750 calorie medium-fat evening meal.
  Arms: Sequence 4
Drug: Sequence 4 - Treatment E: Immediate Release Pregabalin — 300 mg IR capsule administered in the evening in the fasted state.
  Arms: Sequence 4

SUMMARY:
This study is an open-label, single dose, randomized, 5-period, 5-treatment, 4-sequence cross-over with a fixed 5th treatment arm. Subjects will receive in a randomized sequence a 330 mg CR tablet with fast in vitro dissolution rate, a 330 mg CR tablet with slow in vitro dissolution rate, a heavier 330 mg CR tablet with fast in vitro dissolution rate or a 330 mg market image reference CR tablet. Subjects will receive a 300mg IR formulation in the 5th period to to estimate and compare the % of dose absorbed versus time profile for the three CR prototype tablets and the CR reference tablet.

ELIGIBILITY:
Inclusion Criteria:

* Subject eligibility should be reviewed and documented by an appropriately qualified member of the investigator's study team before subjects are included in the study.
* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:
* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of febrile illness within 5 days prior to the first dose of study medication.
* Subjects with an estimated creatinine clearance (CLcr) <60 mL/min derived using the method of Cockcroft and Gault1.
* Any condition possibly affecting drug absorption (eg, gastrectomy, irritable bowel syndrome).
* A positive urine drug screen.
* Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from at least 14 days (for nonhormonal methods) or approximately 3 months (for hormonal contraception) prior to the first dose of study medication and for 28 days after the last dose of study medication.
* Use of prescription (other than oral, transdermal, intrauterine, implanted, or injected contraceptives or hormone replacement therapy) or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued at least 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to pregabalin, gabapentin, or other alpha 2 delta ligands.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Previous participation in a study involving pregabalin.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects with active suicidal ideation or suicidal behavior within 1 year prior to Screening as determined through the use of the C-SSRS (Columbia-Suicide Severity Rating Scale) or active ideation identified at Screening or on Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero extrapolated to infinite time (AUClast) | predose to 48hr post dose
Area under plasma concentration-time profile from time zero to time of last quantifiable concentration (AUCinf) | predose to 48hr post dose
Maximum observed concentration within dosing interval (Cmax) | predose to 48hr post dose
Time for Cmax Tmax | predose to 48hr post dose
Terminal half-life (t1/2) | predose to 48hr post dose
Safety endpoints will be evaluated by comparing the incidence and severity of AEs for each of the formulations evaluated | predose to 48hr post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081286